CLINICAL TRIAL: NCT06589999
Title: Detection of Spinal Cord Lesions Using the MP2RAGE Sequence in Inflammatory Diseases of the Neuraxis
Acronym: SCOUT-MS
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2024_2
Record Dates: First submitted 2024-08-02; First posted 2024-09-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients presenting to the imaging department in the context of inflammatory neuraxial disease
  Interventions: Diagnostic Test: MP2RAGE sequence

INTERVENTIONS:
Diagnostic Test: MP2RAGE sequence — Addition of MRI sequence MP2RAGE

SUMMARY:
Since the last revision of the MRI guidelines in multiple sclerosis (MS, MAGNIMS) and the McDonald criteria in 2017, all spinal cord lesions must be counted to increase the sensitivity and specificity of the diagnosis of MS. Focal lesions of the spinal cord are more frequently located in the cervical segments than in the lower segments of the spinal cord and occupy the lateral and posterior columns, although the central grey matter may not be spared. Cervical involvement is difficult to study because of the small size of the lesions and the loss of signal in the cervical region. As a result, the detection of cervical lesions on MRI is sub-optimal.

In this context, standardised acquisition protocols have been proposed.

For MRI of the spinal cord, at least two of the following sagittal sequences are recommended: T2, STIR, double inversion recovery, T1 with gadolinium injection, and/or T2 axial acquisitions.

Recently, our team validated the superiority of 3D PSIR and 3D FGAPSIR sequences, which offer better detection performance than T2 and STIR on 3 Tesla MRI.

Other studies have also shown the contribution of the MP2RAGE sequence to the detection of spinal cord lesions in MS, compared with the set of sequences classically recommended. The MP2RAGE sequence is a T1 sequence, which creates a composite image, limiting field inhomogeneity bias while providing a quantitative T1 map. It has recently been optimised for the spinal cord, and has been only minimally evaluated in the context of MS.

The aim of this study is to evaluate the effectiveness of the MP2RAGE sequence in comparison with the set of conventional sequences recommended for the detection of spinal cord lesions in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years
* scheduled to undergo 1.5T or 3T MRI of the spinal cord as part of an initial assessment or reassessment of inflammatory neuraxial disease.
* Express consent to participate in the study
* Member or beneficiary of a social security scheme

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant women
* Absolute or relative contraindication to 1.5T or 3T MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be offered prospectively to patients presenting to the imaging department for a 1.5T or 3T MRI scan for spinal cord exploration, in the context of inflammatory involvement of the neuraxis.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
In patients with inflammatory neuraxial disease, estimate the number of cervical lesions detected with the MP2RAGE sequence that were not detected with the recommended standard set. | Day 0
  The images will be reviewed by two radiologists who will be blinded to each other and who will each estimate the number of lesions detected on the images obtained with each of the sequences. Images from the same patient (standard set and MP2RAGE) will not be read at the same time.
  Readers will be instructed not to validate a lesion that is too difficult to see, but only those that are true lesions a priori.
  In the event of disagreement between the two radiologists, a consensus will be sought with a third reader.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Fondation Adolphe de Rothschild, Paris, France